CLINICAL TRIAL: NCT00081692
Title: Longitudinal Cardiac Outcomes and Body Composition
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1248; R01HL072838-05 (NIH)
Record Dates: First submitted 2004-04-19; First posted 2004-04-21 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Only receiving data
Oversight: Data Monitoring Committee: No

SUMMARY:
To relate cardiac structure and blood pressure (BP) elevation in adults to childhood BP and body size and composition.

DETAILED DESCRIPTION:
BACKGROUND:

To describe growth events adequately, long-term serial data with frequent measurements at appropriate ages are necessary. The study uses the Fels Longitudinal Study. In the Fels Longitudinal Study, data collection begins at birth, and all children are scheduled for measurements semiannually, on their birthdays and half birthdays, until the age of 18 years, after which they are scheduled every 2 years. The Fels study is unique with a rich 70-year history of ongoing serial data collection enabling the analysis of relationships of variables collected in childhood to cardiovascular risk factors well into late adulthood.

DESIGN NARRATIVE:

The study will link adult cardiac structure and hemodynamic function with long-term serial childhood data for body size, body composition and blood pressure. To address this goal, 685 adult white active participants in the Fels Longitudinal Study, 352 men and 333 women 20 to 70 years of age, will be studied. These adults were selected based on the availability of serial body size data from 2 to 18 years and serial body composition data from 8 to 18 years. Echo cardiographic data for cardiac structure and hemodynamic parameters will be collected from these 685 adults using well defined procedures with a well established quality control and assurance program. The availability of the long-term childhood records of these Fels participants for body size and composition provides a unique opportunity to relate childhood data to subsequent adult data for cardiac structure and blood pressure. The innovative longitudinal statistical analysis used will include covariates such as age, gender, birth year for secular trend, adulthood lifestyle (smoking, alcohol consumption, and physical activity), adult body size and composition, menopause, and medical condition and medication use. The analysis of the hypotheses in this study links cardiac structure and hemodynamic parameters in adulthood to childhood growth and body composition. Such linkages will reveal how various growth and body composition profiles and patterns during childhood can lead either to pathological or to healthy cardiac structure and hemodynamic parameters in adulthood. Understanding adult cardiac outcomes in response to changes in fat and fat-free mass from childhood into adulthood will provide important clues about potential physiologic mechanisms underlying the observed changes in body mass index (BMI). Elucidating adverse relationships through such a linkage can lead to the early identification of children at high risk for adult cardiovascular disease. This investigation will relate direct measures of body composition to adult cardiac structure and hemodynamic parameters.

ELIGIBILITY:
No eligibility criteria

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Echocardiographic measurements were made in 437 male and 492 female adults in the Fels Longitudinal Study who had serial measurements of body composition made and recorded as children. The selection criteria include participants who have at least 10 serial anthropometric visits between 2 and 20 years of age. The anthropometric measurements include weight and height for computation of BMI and blood pressure. Approximately one-half of the sample is 50 years and older.
Sampling Method: Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Established and validated the echocardiographic protocol that was used to generate the serial data on cardiac structure and function in 723 adults in the FLS population . | 1929-2009
  Investigators are currently finishing an investigation of racial divergence in cardiac structure, cardiac function and blood pressure in relationship to child growth from 9 to 18 years in 700 women who were participants in the National Growth and Health Study participants. Preliminary results show that women who were overweight during childhood (25 ≤ BMI < 30 kg/m2) had a significantly larger LVM and elevated systolic blood pressure (SBP) at age 22 years than women who were not overweight during childhood. Women who had elevated SBP during childhood had a significantly larger LVM and elevated SBP at age 22 years than women who did not have elevated SBP values during childhood.

CONTACTS AND LOCATIONS:
Overall Officials: Shumei Sun, PhD, Principal Investigator — Virginia Commonwealth University

REFERENCES:
- [Result] Sabo RT, Lu Z, Daniels S, Sun SS. Serial childhood BMI and associations with adult hypertension and obesity: the Fels Longitudinal Study. Obesity (Silver Spring). 2012 Aug;20(8):1741-3. doi: 10.1038/oby.2012.58. Epub 2012 Mar 8. PMID 22402734
- [Result] Sabo RT, Lu Z, Daniels S, Sun SS. Relationships between serial childhood adiposity measures and adult blood pressure: The Fels longitudinal study. Am J Hum Biol. 2010 Nov-Dec;22(6):830-5. doi: 10.1002/ajhb.21091. PMID 20865760